CLINICAL TRIAL: NCT06432959
Title: Incorporating Positive Affect Into Cognitive Behavioral Therapy for Depression and Dialectical Behavior Therapy for Borderline Personality Disorder and Severe Emotion Dysregulation
Brief Title: Incorporating Positive Affect Promoting Activities Into Cognitive Behavioral Therapies
Acronym: PAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Cheavens, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022B0257
Record Dates: First submitted 2023-03-22; First posted 2024-05-29 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Depression; Borderline Personality Disorder; Emotion Regulation
MeSH Terms: conditions — Depression; Borderline Personality Disorder; Emotional Regulation | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Masking Description: Participants will be randomized to treatment as usual (i.e., CBT or DBT) or treatment-as-usual plus positive affect promoting activities (i.e., CBT with PAPA, DBT with PAPA). Randomization will occur within clinic (i.e., one clinic provides CBT, the other provides DBT). In the clinic providing CBT for depression, a total of 50 participants will be randomized (25 each to CBT or CBT with PAPA). In the clinic providing DBT, 40 participants will be randomized (20 each to CBT or CBT with PAPA). Given the treatments under investigation, neither the interventionist nor the participant could be kept unaware of condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Participants in the TAU arm will receive either Cognitive Behavioral Therapy (CBT) or Dialectical Behavior Therapy (DBT), depending on eligibility. CBT will be twice weekly sessions for the first four weeks. From week 4 to week 8, the therapist and client will collaboratively decide whether to have once or twice weekly sessions. From week 8 to week 12, sessions will be weekly. Acute treatment will end after 12 weeks. In DBT, individual sessions will be approximately one hour per week, with optional additional or longer sessions available if deemed clinically necessary, and group sessions will be scheduled for two hours once per week.
  Interventions: Behavioral: Psychotherapy
- TAU + Positive Affect Promoting Activities (Experimental): Those assigned to the PAPA condition will also receive either CBT or DBT, as described above, and additionally will be asked to participate in positive affective promoting activities. In session positive affective promoting activities are to be provided once per week for the first four weeks of treatment and up to once per session for the remaining sessions. Clients will also be encouraged to utilize positive affect promoting activities between sessions.
  Interventions: Behavioral: Psychotherapy, Positive Affect Promoting Activities; Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy, Positive Affect Promoting Activities — The specific activities that constitute the positive affect interventions will be determined by the therapist and participant collaboratively. Some examples of positive affect promoting activities are:
  * Watch videos of animals and babies
  * Eat a piece of candy
  * Recall and describe a past positive experience
  * Describe the positive attributes of the participant
  * Engage in gratitude practice
  * Do something nice for someone
  The in-session positive affect activities will last approximately five minutes. For the first four weeks, the positive affect activities will be completed at the beginning of the session. After that, therapists will look for opportunities to incorporate positive affect activities at "stuck points" or before learning a new skill in-session. Additionally, therapists will work with participants to identify ways in which the participants can incorporate positive affect activities into their lives between sessions.
  Arms: TAU + Positive Affect Promoting Activities
Behavioral: Psychotherapy — Meet with treatment providers individually or in group to learn skills to address symptoms associated with depression and emotion dysregulation

SUMMARY:
In this study, the investigators will test whether the incorporation of positive affect promoting activities in treatment sessions improves outcomes in the context of CBT for depression and DBT for problems of emotion dysregulation. In clinics focused on each of these treatments, the investigators will evaluate these treatments with and without the addition of positive affect promoting activities.

DETAILED DESCRIPTION:
The investigators will randomize participants to treatment with or without positive affect promoting activities in two samples of adults with emotional disorders participating in a form of cognitive behavioral therapy. One sample will be drawn from a clinic providing CBT for depression and the other will be drawn from a clinic providing dialectical behavior therapy.

This study is a two-clinic randomized clinical trial. Eligible participants will be randomized to standard treatment or standard treatment + positive affect promoting activities. A total of 50 participants (25 per condition) will be randomized in a clinic providing CBT for depression. A total of 40 (20 per condition) will be randomized in a clinic providing CBT for problems of emotion dysregulation. Treatment will be provided over 12 weeks in the CBT for depression clinic sample and 24 weeks in the DBT clinic sample. At pre-treatment, 4-weeks, and 12-weeks, participants will complete symptoms measures in addition to measures of diagnosis-relevant processes (e.g., rumination), personality, therapy skills, treatment engagement, and treatment history. Additionally, participants and providers will complete measures before and after each therapy session to assess alliance, engagement, symptoms, skills, and mood. Sessions will be recorded to later code psychotherapy process measures.

CBT. Clients will participate in a course of CBT for depression. CBT consists of a series of structured, collaborative sessions with a focus on promoting behavioral activation and helping patients to re-evaluate unduly negative views (e.g., "I am worthless"). Treatment will be informed by the primary treatment manual for CBT of depression. Additional cognitive-behavioral treatment procedures for co-occurring conditions may be used as judged appropriate. Study personnel will provide treatment and all clinical assessments. Clinical supervision will be provided by a licensed psychologist.

The protocol for CBT will be to have twice weekly sessions for the first four weeks. From week 4 to week 8, the therapist and client will collaboratively decide whether to maintain twice weekly sessions or switch to once weekly sessions. From week 8 to week 12, sessions will be weekly. Acute treatment will end after 12 weeks. Clients will have the option of consulting with their therapist or another therapist (which would be likely when a therapist is no longer providing treatment for the study) for up to two booster sessions in the six months following their 12-week acute treatment period.

DBT. Clients will participate in a six-month (24 to 26-week) course of DBT. DBT consists of weekly individual and group psychotherapy sessions that focus on enhancing skills in mindfulness, interpersonal effectiveness, emotion regulation, and distress tolerance. Individual sessions will be approximately one hour per week, with optional additional or longer sessions available if deemed clinically necessary, and group sessions will be scheduled for two hours once per week. At study end, participants who wish to continue treatment will be provided with referrals in the community or in the clinic, if therapists are available.

Study personnel will provide treatment and all clinical assessments. Clinical supervision will be provided by a licensed psychologist. Recent evidence suggests that 6-months of DBT results in similar outcomes when compared to 12-months of DBT. The research group has demonstrated that DBT delivered in a training clinic with this protocol is associated with gains in the domains targeted in the treatment.

Positive Affect Promoting Activities Participants will be randomized to either the Positive Affect Promotion Activities (PAPA) condition or the treatment-as-usual (TAU) condition. Patients in the TAU condition will receive either CBT or DBT as described above. Those assigned to the PAPA condition will also receive either CBT or DBT, as described above, and additionally will be asked to participate in a positive affective promoting activities once per week for the first four weeks of treatment and up to once per session for the remaining sessions. Following the first four weeks, therapists will work with clients to identify occasions to use positive affect induction procedures as part of between session coping strategies and as method to facilitate subsequent use of additional strategies (both in session and between sessions).

The specific activities that constitute the positive affect interventions will be determined by the therapist and participant collaboratively. Given that there are individual differences in the ways that people appraise various stimuli, it is important to be flexible in determining what might be an effective positive affect promoting activity for each participant. Some examples of positive affect promoting activities that might be incorporated into therapy sessions or between therapy sessions include:

* Watch videos of animals (e.g., dogs, pandas, penguins) and babies (e.g., laughing, discovering)
* Eat a piece of candy
* Recall and describe a past positive experience (e.g., talk about success, interest / goal pursuit)
* Describe the positive attributes of the participant
* Engage in gratitude practice
* Do something nice for someone (e.g., write thank you notes for deployed troops, notes of encouragement for children in the hospital, volunteer)
* Listen to music
* Draw or create
* Practice mindfulness, including loving kindness meditations
* Take a walk or dance
* Watch clips of comedians
* Go outside and sit in the sun
* View pictures of loved ones/animals

The in-session positive affect activities will last approximately five minutes. For the first four weeks, the positive affect activities will be completed at the beginning of the session. After that, therapists will look for opportunities to incorporate positive affect activities at "stuck points" or before learning a new skill in-session. Additionally, therapists will work with participants to identify ways in which the participants can incorporate positive affect activities into their lives between sessions. Participants and therapists will work together to identify activities that reliably lead to feeling joy, curiosity, pride, or love, for example. Then, therapists will work with participants to find opportunities to engage in these activities to help motivate themselves to engage in difficult tasks, learn new things, or regulate their emotions.

ELIGIBILITY:
Clinic-specific inclusion criteria are as follows. For the clinic providing CBT for depression, participants must meet criteria for a diagnosis of major depressive disorder according to Diagnostic and Statistical Manual-5 (DSM-5). They must also be able to attend in-person sessions or have access to a reliable internet connection to participate in virtual sessions.

For the clinic providing DBT, participants must evidence severe emotion dysregulation defined as (1) meeting criteria for borderline personality disorder (BPD) or (2) elevated indicators of borderline personality pathology defined as average scores of 1.5 on the Personality Inventory for DSM-5 (PID-5) Negative Affectivity scale and 1.25 on the Antagonism scale and/or 1.25 on the Disinhibition scale. They must also be willing and able to attend in-person sessions.

Across both clinics, the following inclusion and exclusion criteria will be applied:

Inclusion Criteria:

1. 18 years old or older
2. residence in the state of Ohio
3. able and willing to give informed consent

Exclusion Criteria:

1. current or past diagnosis of bipolar disorder or a psychotic disorder
2. presence of a psychiatric disorder other than Major Depressive Disorder (MDD) or BPD, if it constitutes the predominant aspect of the clinical presentation and if it requires treatment other than that being offered (including substance use disorders involving heroin, cocaine, and methamphetamine deemed inappropriate at pre-screening)
3. currently participating in a psychosocial treatment for an emotional disorder, including any individual psychotherapy
4. if on psychiatric medication, no changes to medication regimen (drugs or dosage) in the past month and no intention to modify medication regimen for the next 12 weeks
5. clear indication of secondary gain (e.g., court-ordered treatment)
6. current suicide risk of medical instability (e.g., low weight) to preclude treatment on an outpatient basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Weekly Change in Quick Inventory of Depressive Symptoms, Self-Report | weekly over 12 weeks
  16 item self-report assessment of symptoms of depression with each item scored on a 0-3 scale. Higher scores indicate more severe symptoms of depression.
Weekly Change in Positive and Negative Affect Schedule | weekly over 12 weeks
  20 item self-rated assessment of positive and negative affect in the moment with each item scored on a 1-9 scale. Higher scores reflect higher levels of affect.

SECONDARY OUTCOMES:
Weekly Change in Impressions of Skills Scale | weekly over 12 weeks
  Measure developed for this study to assess use, understanding, and confidence in using therapy skills. There are seven items, each rated on a scale of 1-7. Higher scores indicate that the participant more fully understood the skills taught in session and is confident they will be able to use the skills outside of session.
Change in Credibility/Expectancy Questionnaire | 4 weeks
  6 item questionnaire used to assess expectations of treatment with four items measuring confidence or expectations for the treatment (scored 1 - 9) and two items assessing anticipated improvement in symptoms (scored 0 - 100%). Higher scores reflect more confidence and expected improvement.
Weekly Change in Working Alliance Inventory | weekly for 12 weeks
  Completed by both participants and providers to assess quality of the therapeutic relationship. This scale has 12-items and each is scored 0 - 6. Higher scores reflect a better therapeutic relationship.

OTHER OUTCOMES:
Change in Personality Assessment Inventory - Borderline Personality Disorder Subscale | 12 weeks
  24-item self-report assessment of BPD features, will be used as an outcome measure for those in the DBT clinic. Each item is rated as "false," "slightly true," "mainly true," or "very true." Higher scores suggest more severe BPD features.
Change in Personality Inventory for DSM-5 - Faceted Brief Form | 12 weeks
  100 item self-report measure of personality traits, including specifically for this study antagonism, neuroticism, and disinhibition. Each item is rated on a scale from 0 - 3 with higher scores reflecting more of a given trait.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will consider requests for data sharing, pending approval from our Institutional Review Board (IRB).
  Note: Individual participant data (IPD).

DOCUMENTS (2):
  • Informed Consent Form: ICF for Participants in the DBT Clinic (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT06432959/ICF_000.pdf
  • Informed Consent Form: ICF for Participants in the Depression Clinic (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT06432959/ICF_001.pdf